CLINICAL TRIAL: NCT03095963
Title: Effects of Probiotics Assumption on Serum Thyroid Hormone and TSH Levels in Hypothyroid Patients on Levothyroxine Treatment
Brief Title: Interaction Between Levothyroxine and Probiotics in Hypothyroid Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Modena (Other)
Responsible Party: Principal Investigator, Manuela Simoni, Director of Unit of Endocrinology, Department of Medicine, Endocrinology, Metabolism and Geriatrics, Azienda Ospedaliero-Universitaria of Modena, Modena, Italy, Azienda USL Modena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Levothyroxine and Probiotics
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): The study group took a mixture of highly charged Lactobacilli and Bifidobacteria (VSL#3®) in addition to levothyroxine
  Interventions: Other: a mixture of highly charged Lactobacilli and Bifidobacteria (VSL#3®); Drug: levothyroxin
- Levothyroxine (Active Comparator): The control group took levothyroxine only
  Interventions: Drug: levothyroxin

INTERVENTIONS:
Other: a mixture of highly charged Lactobacilli and Bifidobacteria (VSL#3®) — Patients assigned to the study group took the probiotic supplement VSL#3® for two months, in addition to levothyroxine
  Arms: Probiotics
Drug: levothyroxin — replacement therapy for hypothyroidism

SUMMARY:
A prospective, randomized, single-blind, controlled, investigator-started clinical trial was carried out. Patients with primary hypothyroidism were randomly assigned to the study (VSL#3®+ LT4) and the control group (LT4). A two months treatment phase was followed by two months of follow-up. Clinical examination, blood tests for thyroid function and for peripheral tissue markers of thyroid hormones effect were performed monthly for 4 months. LT4 dose adjustments were performed during the study when necessary.

DETAILED DESCRIPTION:
Consecutive patients on LT4 replacement therapy attending the Endocrinology Unit of Modena (Italy) were screened. According to inclusion and exclusion criteria, eighty participants were enrolled and randomized in study or control group. The random allocation sequence was generated using 'Statistical Package for the Social Sciences' software for Macintosh (SPSS) considering a 1:1 ratio by the statistician of the Unit. Clinicians evaluating and enrolling patients were blinded to the randomization list. The study design provided a monthly visit for a 4 months overall time-frame. Patients assigned to the study group took the probiotic supplement VSL#3® for two months, followed by a two months period of follow-up. Study group patients were taught to assume the probiotic supplement at least two hours after LT4 administration, to dissolve it in a cold beverage and to store it in a refrigerator (2°-8°C) in order to preserve bacteria load. The study design was single-blind since only the clinician was aware of the allocation. The VSL#3® administration was provided by nurses. Participants were invited to return all used and unused sachets to count the number of opened sachets per the number of treatment days.

All patients underwent five visits (baseline, visit 1, 2, 3 and 4) in which anthropometrical evaluation (weight and height) and hormonal function assessment were performed. A blood sample was taken in the morning at each visit, on empty stomach and before LT4 ingestion. In occurrence of hormonal alteration, LT4 daily dose was adjusted according to clinical guidelines. At baseline, visit 2 and visit 4, patients underwent clinical examination with heart rate and blood pressure evaluation. During each visit, the following data were collected: probiotic assumption, sex, age, hypothyroidism aetiology, LT4 formulation dose and brand, body mass index (BMI), body surface area (BSA), systolic blood pressure, diastolic blood pressure, heart rate, TSH, fT4, fT3 and any possible LT4 posology adjustment. All the clinical data have been further databased.

ELIGIBILITY:
Inclusion Criteria:

* primary hypothyroidism on LT4 replacement therapy
* TSH, fT3 and fT4 in the normal range
* stable LT4 dosage during the previous six months before enrolment
* Caucasian ethnicity

Exclusion Criteria:

* total thyroidectomy for thyroid carcinoma
* high fiber diet
* intestinal malabsorption (e.g. bariatric surgery, inflammatory bowel diseases, coeliac disease)
* ongoing therapies interfering with LT4 absorption and/or metabolism (i.e. aluminium-containing antacids, sucralfate, proton pump inhibitors, calcium carbonate, raloxifene, bile acids sequestrants and ferrous sulfate)
* antibiotics treatment in the previous six months before enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01-01; Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
differences in thyroid-stimulating hormone (TSH) serum levels comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of thyroid-stimulating hormone (TSH) - unit of measure: microIU/mL, normal range: 0.35-4.94

SECONDARY OUTCOMES:
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of total cholesterol (CH) - unit of measure: mg/dL, normal range: <200
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of sex hormone-binding globulin (SHBG) - unit of measure: nmol/L, normal range: males 13.5-71.4, females 19.8-155.2
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of ferritin - unit of measure: ng/mL, normal range: 25-400
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of creatine phosphokinase (CPK) - unit of measure: U/L, normal range: 10-71
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of myoglobin - unit of measure: ng/mL, normal range: 15-106
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of osteocalcin - unit of measure: ng/mL, normal range: 4.6-65.4
differences in peripheral tissue markers of thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of angiotensin-converting enzyme (ACE) - unit of measure: U/L, normal range: 8-52
differences in thyroid hormones by biochemical assays comparing study group and controls | Through study completion, an average of 4 months
  measurement of serum levels of free triiodothyronine (fT3) - unit of measure: pg/mL, normal range: 1.7-3.7; measurement of serum levels of free thyroxine (fT4) - unit of measure: pg/mL, normal range: 7-15

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spaggiari G, Brigante G, De Vincentis S, Cattini U, Roli L, De Santis MC, Baraldi E, Tagliavini S, Varani M, Trenti T, Rochira V, Simoni M, Santi D. Probiotics Ingestion Does Not Directly Affect Thyroid Hormonal Parameters in Hypothyroid Patients on Levothyroxine Treatment. Front Endocrinol (Lausanne). 2017 Nov 14;8:316. doi: 10.3389/fendo.2017.00316. eCollection 2017. PMID 29184537